CLINICAL TRIAL: NCT03300362
Title: A Phase IIb Study to Determine the Safety and Efficacy of Candidate INfluenza Vaccine MVA-NP+M1 in Combination With Licensed InaCTivated inflUenza Vaccine in adultS Aged 65 Years and Above
Brief Title: Improved Novel VaccIne CombinaTion InflUenza Study
Acronym: INVICTUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change to recommended season flu vaccine in UK
Sponsor: Barinthus Biotherapeutics (Industry)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLU007 INVICTUS
Record Dates: First submitted 2017-09-26; First posted 2017-10-03 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Investigators recording clinical outcomes will also be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seasonal influenza & MVA-NP+M1 (Experimental): Two vaccinations will be administered: Seasonal influenza vaccine & MVA-NP+M1
  Interventions: Drug: Seasonal influenza vaccine; Drug: MVA-NP+M1
- Seasonal influenza & saline placebo (Placebo Comparator): Two vaccinations will be administered: Seasonal influenza vaccine & sodium chloride
  Interventions: Drug: Seasonal influenza vaccine; Drug: Sodium chloride

INTERVENTIONS:
Drug: Seasonal influenza vaccine — Seasonal influenza vaccine
  Other Names: Quadrivalent Influenza Vaccine
Drug: MVA-NP+M1 — Trial vaccine
  Arms: Seasonal influenza & MVA-NP+M1
Drug: Sodium chloride — Saline placebo
  Arms: Seasonal influenza & saline placebo

SUMMARY:
A Phase IIb randomised, participant-blinded, placebo-controlled, multi-centre phase IIb efficacy study in 2030 volunteers aged 65 and over. The study will assess the safety and efficacy of the co-administration of a viral vectored vaccine, MVA- NP+M1, and the annual recommended licensed inactivated influenza vaccine (IIV). Within the main cohort 100 participants will be recruited to an immunology sub-cohort.

DETAILED DESCRIPTION:
The efficacy of current seasonal influenza vaccines is limited in the face of antigenic mismatch between circulating viral strains and those in the given vaccine. Additionally vaccination in older adults, a major target group for vaccination, prevents laboratory-confirmed influenza in only 30-40% compared to 70-90% in young adults. The hypothesis in this Phase IIb efficacy study is that a new vaccine MVA-NP+M1 with licensed inactivated influenza vaccine (IIV) in the older age group will be able to induce immune responses that protect individuals against influenza illness, severity of symptoms and reduce viral shedding, thereby increasing the protection conferred by seasonal influenza vaccine alone. A total of 2030 participants who are 65 years of age or over and eligible for annual seasonal influenza vaccination and provide informed consent will be recruited to the study. Potential volunteers will be mailed an invitation to take part by their GPs or recruited by local advertisements. Participants will be randomised to receive either MVA- NP+M1 with licensed IIV or saline placebo with licensed IIV. In the first 28 days after vaccination, participants will record adverse events using an electronic or paper diary. The participants will be contacted by telephone 1 day and 7 days post-vaccination to enquire about any serious adverse events and support follow up. During influenza season participants will record weekly whether or not they have had an influenza like illness (ILI). For every ILI episode experienced, the participants will record the severity of their symptoms daily. Among the participants, a total of 100 volunteers (50 in each group) will be recruited into an immunology sub-cohort. They will have blood samples collected on the day of vaccination, 1 week, 3 weeks and 26 weeks post-vaccination for monitoring of laboratory adverse events and immunogenicity purposes.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer is willing and has capacity to provide written informed consent for participation in the trial (in the Investigator's opinion).
* Male or female adults, aged 65 years and above
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* Eligible to receive seasonal influenza vaccine

Exclusion Criteria:

* Any history of anaphylaxis in reaction to vaccination or history of allergic reactions likely to be exacerbated by any component of the vaccine (e.g. egg allergy)
* Ongoing terminal illness with a life expectancy estimated to be approximately <6 months.
* Continuous use of oral anticoagulants, such as coumarins and related anticoagulants (i.e. warfarin) or novel oral anticoagulants (i.e. apixaban, rivaroxaban, dabigatran and edoxaban)
* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigators, would either put the volunteer at risk because of participation in the study, or may influence the result of the study
* Participation in another clinical trial of an investigational medicinal product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data
* Receipt of annual seasonal influenza vaccine prior to enrolment (for the same influenza season volunteers are recruited in)
* Not willing to comply with study procedures

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 862 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Number of days with moderate or severe influenza-like symptoms | 6-7 months
  Throughout the influenza season, self-reported symptoms recorded using electronic or paper diaries

SECONDARY OUTCOMES:
Incidence of influenza-like-illness | 6-7 months
  Throughout the influenza season, self-reported symptoms recorded using electronic or paper diaries
Severity of influenza-like symptoms | 6-7 months
  Throughout the influenza season, self-reported symptoms recorded using electronic or paper diaries
Duration of influenza-like-illnes | 6-7 months
  Throughout the influenza season, self-reported symptoms recorded using electronic or paper diaries
Occurrence of GP consultations from respiratory illness | 6-7 months
  Throughout the influenza season - self-reported and Medical Records
Occurrence of hospitalisations and deaths due to respiratory illness | 6-7 months
  Throughout the influenza season - self-reported and Medical Records
Occurrence of solicited local and systemic reactogenicity signs and symptoms for 7 days following vaccination | Day 0-7
  Self-reported symptoms recorded using electronic or paper diaries
Occurrence of serious adverse events during the whole study duration | 6-7 months
  Telephone calls on Day 1-3, day 7-9 and every 3-4 weeks throughout volunteers' participation in the trial
Occurrence of unsolicited adverse events for 28 days following vaccination | Day 0-28
  Self-reported symptoms recorded using electronic or paper diaries
Frequency of influenza-specific T-cells measured by IFNg ELISpot | 6-7 months
  To assess the immunogenicity of MVA-NP+M1 in combination with the recommended licensed inactivated influenza vaccine in adults aged 65 years and above
Geometric mean titre of influenza-specific neutralising antibodies | 6-7 months
  To assess the immunogenicity of MVA-NP+M1 in combination with the recommended licensed inactivated influenza vaccine in adults aged 65 years and above
Breadth of influenza-specific T-cells and antibodies | 6-7 months
  To assess the immunogenicity of MVA-NP+M1 in combination with the recommended licensed inactivated influenza vaccine in adults aged 65 years and above

OTHER OUTCOMES:
Estimated frequency of influenza infection using historical data on the proportion of ILIs that is caused by influenza virus infection. | 6-7 months
  To explore novel clinical endpoints for future Phase III efficacy trials of influenza vaccines

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Butler, Principal Investigator — University of Sussex
Locations (5):
- United Kingdom (5):
  - The Boathouse Surgery, Pangbourne, Berkshire
  - Wokingham Medical Centre, Wokingham, Berkshire
  - Bicester Health Centre, Bicester, Oxfordshire
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM, Oxford, Oxfordshire
  - Windrush Health Centre, Witney, Oxfordshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swayze H, Allen J, Folegatti P, Yu LM, Gilbert S, Hill A, Ellis C, Butler CC. A phase IIb study to determine the safety and efficacy of candidate INfluenza Vaccine MVA-NP+M1 in combination with licensed Ina CTivated infl Uenza vaccine in adult S aged 65 years and above (INVICTUS): a study protocol. F1000Res. 2019 May 23;8:719. doi: 10.12688/f1000research.19090.1. eCollection 2019. PMID 32089822